CLINICAL TRIAL: NCT03858946
Title: Ligament Reconstruction Interpositions Arthroplasty Modo Weilby Versus Simple Trapeziectomy for Primary Thumb Carpometacarpal Osteoarthritis
Brief Title: Ligament Reconstruction Weilby vs Simple Trapeziectomy
Acronym: WEILBY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Carsten Jensen, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-20170041
Record Dates: First submitted 2019-02-22; First posted 2019-03-01 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the TI group, two shame incisions will be performed to mimic those, incisions made during FCR tendon harvesting in the LRTI group. Hence, blinding to treatment allocation of patients, physiotherapists and health care providers will be possible. Furthermore, independent data collectors will be responsible for baseline and follow-up assessments, while all self-reported outcome questionnaires are made available to the patients electronically, and responses entered into a database identified by identification numbers only. The data analyst will be unaware of the treatment allocation as data will be analyzed using recoded identification numbers. An independent person will perform the recoding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple trapeziectomy (Sham Comparator): Simple trapeziectomy with two sham incisions for primary thumb carpometacarpal osteoarthritis
  Interventions: Procedure: Simple trapeziectomy
- Weilby (Experimental): Ligament reconstruction interpositions arthroplasty modo Weilby for primary thumb carpometacarpal osteoarthritis
  Interventions: Procedure: Weilby

INTERVENTIONS:
Procedure: Simple trapeziectomy — A curvilinear incision is made over the base of the 1. metacarpal towards the tendon of the extensor pollicis brevis in the distal part of the anatomical snuffbox. The joint is opened as widely as possible and the trapezium is dissected free in a proximal direction until the articulation with the scaphoid is reached. Then trapezium is removed taking care not to damage tendon of the flexor carpi radialis. The joint capsule is closed and skin sutured in the usual manner. At the completion of the procedure two small shame incision are made (1 cm each) involving only epidermis on the volar aspect of the palm and forearm. Each of them will be closed with one stitch
  Arms: Simple trapeziectomy
Procedure: Weilby — The first part of the surgical procedure is identical to simple trapeziectomy. In addition, the tendon sheath of the first extensor compartment is divided. After this, a strip consisting of approximately one-third of flexor carpi radialis tendon is dissected using two small incisions on the volar aspect of the wrist and distal forearm. The distally based tendon strip is tunneled to its insertion on the second metacarpal bone. Then the strip of tendon is winded around the abductor pollicis longus tendon and the rest of the tendon at least twice, pulling those tendons together into the space created after excision of the trapezium. The tendons are sutured together with non-absorbable sutures while the skin is sutured in the usual manner
  Other Names: Ligament reconstruction interpositions arthroplasty
  Arms: Weilby

SUMMARY:
There is currently no consensus on the best surgical approach for carpometacarpal osteoarthritis treatment. Simple trapeziectomy (TI) or trapeziectomy with ligament reconstruction tendon interposition (LRTI) are both accepted procedures but evidence is lacking. We want to conduct a high quality prospective randomized trial in which preoperative and postoperative objective and subjective outcome measures of both procedures will be compared.

In this trial, investigators compare the Weilby procedure (LRTI) to simple trapeziectomy (TI) with shame incisions in patients with severe trapeziometacarpal osteoarthritis. Investigators hypothesize that TI will be equal to LRTI in terms of both subjective and objective outcome measures

DETAILED DESCRIPTION:
Trapeziometacarpal (TM) osteoarthritis is the second most common location of osteoarthritis in the hand and one of the most common arthritis sites of all joints. The prevalence of isolated radiographic TM joint arthritis is 35% in people older than 55 years. Armstrong et al. reported TM joint arthritis prevalence of 33% in postmenopausal women, of which one third was symptomatic and prevalence of 11% in men older than 55 years. A pathology involving thumb TM joint may lead to functional disability of the entire hand due to pain, weakened pinch/grip strength and decreased thumb opposition. The most common classification system described is Eaton and Litter using 4 stages of thumb TM joint arthritis. The indication for surgical treatment includes pain, TM joint deformity, grip weakness that interfere with daily functions and no response to conservative treatment. A variety of different procedures has been proposed for treatment of TM arthritis. For less severe stages (Eaton-Littler type 1 and 2) operative options include hemi-trapeziectomy, volar ligament reconstruction, thumb metacarpal osteotomy and arthroscopically assisted debridement/synovectomy of the TM joint.For more severe stages (Eaton-Littler type 3 and 4) TM joint arthrodesis, TM primary joint arthroplasty, trapeziectomy alone or combined with use of ligament augmentation.

Limitation of TM joint arthrodesis includes risk of nonunion, decreased thumb motion and degenerative changes to adjacent joints. TM joint arthroplasty leads to fast pain relief, stronger grip function and improved range of motion during short-term postoperative course but long-term risk of implant failure and aseptic loosening has been reported. The aim of trapezial excision is to remove the arthritic TM joint thus reducing pain and maintaining thumb mobility.Several studies have reported excellent results after trapeziectomy.

However, simple excision of the trapezium was criticized for weakening of the thumb, due to instability and proximal migration of the 1. metacarpal. To overcome this issue several surgical technics were described in which trapezium resection is combined with ligament reconstruction tendon interposition (LRTI). Interposition is achieved by placing the rolled-up tendon autograft into the space between the scaphoid and 1. metacarp and stabilization by ligament reconstruction at the base of 1. metacarp. A variety of different LRTI procedures including harvesting of the flexor carpi radialis tendon (FCR), extensor carpi radialis longus tendon (ECRL), abductor pollicis longus tendon (APL) and palmaris have been described.

However, Weilby published in 1988 a method of ligament reconstruction utilizing the half of the width of the flexor carpi radialis tendon (FCR). The strip of the FCR is harvested and coiled around abductor pollicis longus and itself thus restoring metacarpal stability and preventing its subsidence. Today, the Weilby procedure is the most common type of LRTI operations in Denmark. Despite of Weilby's widespread use there is lack of evidence for the superiority of the procedure over simple trapeziectomy in terms of pain reduction, changes in range of motion and muscle strength and studies describes adverse effects of LRTI procedures, which include FCR tendon ruptures or adhesions, scar tenderness, sensory changes, neuromas, complex regional pain syndrome and wound infections.

In contrast, fewer complications and adverse effects have been reported after simple trapeziectomy. In summary, there is insufficient evidence which technique confers a benefit over another technique in terms of pain, physical function, strength and complications. To the investigators knowledge, no trial exist that compared LRTI to simple trapeziectomy with sham surgery.

ELIGIBILITY:
Inclusion Criteria:

Primary carpometacarpal osteoarthritis Unresponsive to conservative treatment Ability to read and/or understand Danish

Exclusion Criteria:

Rheumatoid arthritis or other types of inflammatory arthritis Previous surgery of the hand TM joint arthritis stage Eaton Litter 1 or 2 TM arthritis due to fracture/dislocation Congenital thumb disorders Other types of surgery in addition to trapeziectomy / Weilby

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in physical function and symptoms | Change from baseline at 12 months
  The shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH) with 11 items measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. Scores range from 0-100. A higher score indicates greater disability.

SECONDARY OUTCOMES:
Change in Self-reported pain | Change from baseline at 12 months
  Visual Analog Scale (VAS). Scores range from 0-100. A higher score indicates more pain.
Change in palmar abduction range of motion | Change from baseline at 12 months
  The range of motion of palmar abduction is assessed. The units of measure is degrees
Change in palmar extension range of motion | Change from baseline at 12 months
  The range of motion of palmar extension (lateral abduction) is assessed. The units of measure is degrees
Change in palmar opposition range of motion | Change from baseline at 12 months
  The range of motion of palmar opposition is assessed. The units of measure is degrees
Change in grip strength | Change from baseline at 12 months
  Isometric Maximal Muscle Strength. The units of measure is Newton

OTHER OUTCOMES:
Adverse events | at 12 months
  A medical audit will be conducted at 12 months post-surgery and information will be obtained by accessing the electronic journal of each participating patient in the trial
Side-effects | at 12 months
  Deep infection, wound bleeding, revision surgery, sensory impairments, swelling and stiffness

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Dept. of Orthopedic Surgery and Traumatology, Kolding Hospital, Denmark, Kolding
  - Division of Hand Surgery, Dept. of Orthopedics and Traumatology, Hospital of Southern Denmark, Sønderborg
  - Division of Hand Surgery, Dept. of Orthopedics, Vejle Hospital, Vejle